CLINICAL TRIAL: NCT01474135
Title: A Double-masked, Randomized, Controlled Study Assessing the Safety and Ocular Hypotensive Efficacy of Two AR 12286/Travoprost Fixed-dose Combination Products Compared to Travatan® Z in Patients With Elevated Intraocular Pressure
Brief Title: AR-12286 Fixed Dose Combination to Lower Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG286-CS201
Record Dates: First submitted 2011-11-11; First posted 2011-11-18 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — AR-12286; Travoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.25% AR-12286/ 0.004% travoprost (Experimental): Fixed dose combination of 0.25% AR-12286 and 0.004% travoprost
  Interventions: Drug: 0.25% AR-12286 / 0.004% travoprost
- 0.5% AR-12286/ 0.004% travoprost (Experimental): Fixed dose combination of 0.5% AR-12286/ 0.004% travoprost
  Interventions: Drug: 0.5% AR-12286, 0.004% travoprost
- 0.004%Travoprost (Active Comparator): Travatan(R) Z(travoprost ophthalmic solution)
  Interventions: Drug: 0.004% Travoprost

INTERVENTIONS:
Drug: 0.25% AR-12286 / 0.004% travoprost
  Arms: 0.25% AR-12286/ 0.004% travoprost
Drug: 0.5% AR-12286, 0.004% travoprost
  Arms: 0.5% AR-12286/ 0.004% travoprost
Drug: 0.004% Travoprost
  Arms: 0.004%Travoprost

SUMMARY:
This is a double-masked, randomized, controlled study assessing the safety and ocular hypotensive efficacy of two AR 12286/travoprost fixed-dose combination products compared to Travatan® Z in patients with elevated intraocular pressure

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout) IOP ≥ 24 mm Hg at 2 eligibility visits (08:00 hr), 2-7 days apart. At second eligibility visit, IOP >22 mmHg at 10:00, 12:00 and 16:00 hrs.
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic (in either eye):

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure. Note: Previous laser peripheral iridotomy is acceptable.
2. Intraocular pressure > 36 mm Hg
3. Known hypersensitivity to travoprost, any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s).
5. Refractive surgery in study eye(s) (e.g., radial keratotomy, PRK, LASIK, etc.).
6. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
7. History or evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 1), or of herpes simplex keratitis
8. Contact lens wear within 30 minutes of instillation of study medication.
9. Ocular medication of any kind within 30 days of Visit 1, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 1) or c) lubricating drops for dry eye (which may be used throughout the study).
10. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (i.e., cup-disc ratio > 0.8).
11. Central corneal thickness greater than 600 µ.
12. Any abnormality preventing reliable applanation tonometry of either eye.

    Systemic:
13. Clinically significant abnormalities in laboratory tests at screening.
14. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
15. Participation in any investigational study within the past 30 days.
16. Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
17. Due to status of nonclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

    -

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mean IOP across subjects within treatment group on Days 1 and 7 at each post-treatment timepoint. | 7 days
  Intraocular pressure

SECONDARY OUTCOMES:
Ocular and systemic safety | 7 days
  Ophthalmic examination and adverse event reports

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - United Medical Research Institute, Inglewood, California
  - Aesthetic Eye Care Institute, Newport Beach, California
  - Bacharach practice, Petaluma, California
  - Centre For Health Care, Poway, California
  - Comprehensive Eye Care, St Louis, Missouri
  - Rochester Ophthalmology Group, Rochester, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Abrams Eye Center, Cleveland, Ohio
  - Cataract & Glaucoma Center, El Paso, Texas